CLINICAL TRIAL: NCT03848065
Title: A Phase I, Double-Blind, Randomized, Multicenter Trial of the Safety,Tolerability, and Immunogenicity of V114 in Healthy Japanese Infants
Brief Title: Safety, Tolerability, and Immunogenicity of V114 in Healthy Japanese Infants (V114-028)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-028; 194669 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal Vaccines
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; Vaccines, Combined

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- V114-SC (Experimental): Infant participants will receive a single 0.5 mL subcutaneous (SC) injection of V114 on Visit 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age). Infant participants will receive a single 0.5 mL SC injection of concomitant study vaccine [Adsorbed Diphtheria-purified Pertussis-tetanus-inactivated polio (Sabin strain) Combined Vaccine (DTaP-IPV) at the same time as V114-SC.
  Interventions: Biological: V114; Biological: Adsorbed Diphtheria-purified Pertussis-tetanus-inactivated polio (Sabin strain) Combined Vaccine (DTaP-IPV)
- V114-IM (Experimental): Infant participants will receive a single 0.5 mL intramuscular (IM) injection of V114 at Visit 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age). Infant participants will receive a single 0.5 mL SC injection of concomitant study vaccine (DTaP-IPV) at the same time as V114-IM.
  Interventions: Biological: V114; Biological: Adsorbed Diphtheria-purified Pertussis-tetanus-inactivated polio (Sabin strain) Combined Vaccine (DTaP-IPV)
- PCV13-SC (Active Comparator): Infant participants will receive a single 0.5 mL subcutaneous (SC) injection of pneumococcal 13-valent conjugate vaccine (PCV13) at Visit 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age). Infant participants will receive a single 0.5 mL SC injection of concomitant study vaccine (DTaP-IPV) at the same time as PCV13-SC.
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine (PCV13); Biological: Adsorbed Diphtheria-purified Pertussis-tetanus-inactivated polio (Sabin strain) Combined Vaccine (DTaP-IPV)

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2 mcg each), serotype 6B (4 mcg) and aluminum phosphate adjuvant (125 mcg) in each 0.5 mL dose.
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114-IM; V114-SC
Biological: Pneumococcal 13-valent Conjugate Vaccine (PCV13) — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F, serotype 6B in each 0.5. mL dose.
  Other Names: PREVNAR 13®
  Arms: PCV13-SC
Biological: Adsorbed Diphtheria-purified Pertussis-tetanus-inactivated polio (Sabin strain) Combined Vaccine (DTaP-IPV) — Single SC dose of 0.5 mL at Visits 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age).

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of V114 administered subcutaneously or intramuscularly in healthy Japanese infants (3 months of age).

ELIGIBILITY:
Inclusion Criteria:

* Healthy (based on a review of medical history and physical examination) based on the clinical judgment of the investigator.
* Male or female 3 months of age inclusive (3 months of age to1 day prior to 4 months of age), at the time of obtaining the informed consent.
* Has a legally acceptable representative who understands the study procedures, alternate treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent.

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease.
* Has a known hypersensitivity to vaccines, any component of the pneumococcal conjugate vaccine or any diphtheria toxoid-containing vaccine
* Has any contraindication to the PCV13 and/or diphtheria, tetanus, acellular pertussis, inactivated polio vaccine (DTaP-IPV) being administered in the study (Refer to approved labeling for contraindication details on PCV13 and DTaPIPV vaccine).
* Has a recent febrile illness (axillary temperature ≥37.5°C) occurring within 72 hours prior to receipt of study vaccine.
* Has a known or suspected impairment of immunological function.
* Has a history of congenital or acquired immunodeficiency.
* Has or his/her mother has a documented hepatitis B surface antigen - positive test.
* Has a known functional or anatomic asplenia.
* Has failure to thrive based on the clinical judgement of the investigator.
* Has thrombocytopenia or a known coagulation disorder contraindicating intramuscular vaccination.
* Has a history of autoimmune disease (including but not limited to systemic lupus erythematosus, antiphospholipid syndrome, Bechet's disease, autoimmune thyroid disease, polymyositis and dermatomyositis, scleroderma, type 1 diabetes mellitus, or other autoimmune disorders).
* Has a known neurologic or cognitive behavioral disorder, including encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive development disorder, and related disorders.
* Has received a dose of any pneumococcal and/or DTaP-IPV vaccine (or vaccine containing any DTaP-IPV component) prior to study entry.
* Meets one or more of the following systemic corticosteroid exclusion criteria: has received systemic corticosteroids (equivalent of ≥ 2 mg/kg total daily dose of prednisone or ≥ 20 mg/d for persons weighing > 10 kg) for ≥ 14 consecutive days and has not completed this course of treatment at least 30 days prior to trial randomization, has received systemic corticosteroids within 14 days prior to the first dose of study vaccine at randomization, and is expected to require systemic corticosteroids (equivalent of ≥ 2 mg/kg total daily dose of prednisone or ≥ 20 mg/d for persons weighing > 10 kg) for ≥ 14 consecutive days within 14 days prior to or 30 days after each vaccination during conduct of the study.(Topical, ophthalmic and inhaled steroids are permitted.)
* Has received other licensed non-live vaccines within the 14 days before receipt of first dose of study vaccine.
* Has received a licensed live virus vaccine within the 28 days before receipt of first dose of study vaccine.
* Has received a blood transfusion or blood products, including immunoglobulins before receipt of first dose of study vaccine.
* Has participated in another clinical study of an investigational product before the beginning or anytime during the duration of the current clinical study. Participants enrolled in observational studies may be included; these will be reviewed on a case by case basis for approval by the Sponsor.
* Has any other reason that, in the opinion of the investigator, may interfere with the evaluation required by the study. (Refer to the Vaccination Guideline in Japan). Reasons may include, but are not limited to, being unable to keep appointments or planning to relocate during the study.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (14):
- Japan (14):
  - Meitetsu Hospital ( Site 2805), Nagoya, Aichi-ken
  - Sotobo Children's Clinic ( Site 2807), Isumi, Chiba
  - Hidaka Children's Clinic ( Site 2803), Dazaifu, Fukuoka
  - Isesaki Municipal Hospital ( Site 2806), Isesaki, Gunma
  - Kawasaki Municipal Hospital ( Site 2802), Kawasaki, Kanagawa
  - Yokosuka Kyosai Hospital ( Site 2804), Yokosuka, Kanagawa
  - Suita Municipal Hospital ( Site 2801), Suita, Osaka
  - Kobayashi Pediatric Clinic ( Site 2816), Fujieda, Shizuoka
  - Nishida Kodomo Clinic ( Site 2811), Tama, Tokyo
  - Fukui Aiiku Hospital ( Site 2809), Fukui
  - Fukui-ken Saiseikai Hospital ( Site 2813), Fukui
  - Kubota Children's Clinic ( Site 2815), Osaka
  - Japanese Red Cross Shizuoka Hospital ( Site 2817), Shizuoka
  - Hosaka Children's Clinic ( Site 2814), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ishihara Y, Kuroki H, Hidaka H, Iwai K, Wan K, Shirakawa M, Sawata M. Safety and immunogenicity of a 15-valent pneumococcal conjugate vaccine in Japanese healthy infants: A Phase I study (V114-028). Hum Vaccin Immunother. 2023 Dec 31;19(1):2180973. doi: 10.1080/21645515.2023.2180973. Epub 2023 Mar 7. PMID 36882898
- [Result] Wan K, Shirakawa M, Sawata M. Descriptive analysis of safety and immunogenicity profiles of a 15-valent pneumococcal conjugate vaccine between subcutaneous and intramuscular administration in a phase 1 study of healthy Japanese infants (V114-028). J Infect Chemother. 2025 Feb;31(2):102539. doi: 10.1016/j.jiac.2024.10.007. Epub 2024 Oct 9. PMID 39384037
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male and female participants of 3 months of age were enrolled in this study.
Groups:
- V114-SC: Infant participants received a single 0.5 mL SC injection of V114 at Visit 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age).
- V114-IM: Infant participants received a single 0.5 mL intramuscular (IM) injection of V114 at Visit 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age).
- PCV13-SC: Infant participants received a single 0.5 mL SC injection of pneumococcal 13-valent conjugate vaccine (PCV13) at Visit 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age).
Period: Overall Study
Arm/Group | V114-SC | V114-IM | PCV13-SC
Started | 44 | 45 | 44
Vaccination 1 | 44 | 45 | 43
Vaccination 2 | 44 | 45 | 43
Vaccination 3 | 44 | 45 | 42
Vaccination 4 | 44 | 44 | 42
Completed | 44 | 44 | 42
Not Completed | 0 | 1 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- V114-IM: Infant participants received a single 0.5 mL IM injection of V114 at Visit 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age).
- PCV13-SC: Infant participants received a single 0.5 mL SC injection of PCV13 at Visit 1, 2, 3 and 5 (approximately 3, 4, 5, and 12 to 15 months of age).
- Total: Total of all reporting groups
Arm/Group | V114-SC | V114-IM | PCV13-SC | Total
Number analyzed (Participants) | 44 | 45 | 44 | 133
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 13.7 (0.8) | 13.9 (1.0) | 13.8 (1.1) | 13.8 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 20 | 58
  Male | 24 | 27 | 24 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 45 | 44 | 133
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 44 | 45 | 44 | 133
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs were injection site erythema (redness), injection site induration (hard lump), injection site pain and injection site swelling.
Time Frame: Day 1 to Day 14 post each vaccination
Population: Analysis population consisted of all randomized participants who received at least one dose of trial vaccine.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-SC | V114-IM | PCV13-SC
Number analyzed (Participants) | 44 | 45 | 43
Percentage of Participants
  Injection Site Erythema (Redness) | 100.0 | 82.2 | 95.3
  Injection Site Induration (Hard Lump) | 90.9 | 77.8 | 100.0
  Injection Site Pain | 38.6 | 28.9 | 41.9
  Injection Site Swelling | 86.4 | 73.3 | 88.4
Statistical Analysis 1: Comparison: V114-SC vs V114-IM; Injection Site Erythema (Redness); Test type: Other; p = 0.004, Miettinen & Nurminen method; Difference in Percentages = 17.8, 95% CI 2-sided [9.0 to 31.4] — Difference = % V114-SC minus % V114-IM
Statistical Analysis 2: Comparison: V114-SC vs PCV13-SC; Injection Site Erythema (Redness); Test type: Other; p = 0.150, Miettinen & Nurminen method; Difference in Percentages = 4.7, 95% CI 2-sided [-3.7 to 15.5] — Difference = % V114-SC minus % PCV13-SC
Statistical Analysis 3: Comparison: V114-IM vs PCV13-SC; Injection Site Erythema (Redness); Test type: Other; p = 0.054, Miettinen & Nurminen method; Difference in Percentages = -13.1, 95% CI 2-sided [-27.6 to 0.2] — Difference = % V114-IM minus % PCV13-SC
Statistical Analysis 4: Comparison: V114-SC vs V114-IM; Injection Site Induration (Hard Lump); Test type: Other; p = 0.091, Miettinen & Nurminen method; Difference in Percentages = 13.1, 95% CI 2-sided [-2.3 to 28.8] — Difference = % V114-SC minus % V114-IM
Statistical Analysis 5: Comparison: V114-SC vs PCV13-SC; Injection Site Induration (Hard Lump); Test type: Other; p = 0.044, Miettinen & Nurminen method; Difference in Percentages = -9.1, 95% CI 2-sided [-21.2 to -0.4] — Difference = % V114-SC minus % PCV13-SC
Statistical Analysis 6: Comparison: V114-IM vs PCV13-SC; Injection Site Induration (Hard Lump); Test type: Other; p = 0.001, Miettinen & Nurminen method; Difference in Percentages = -22.2, 95% CI 2-sided [-36.4 to -12.5] — Difference = % V114-IM minus % PCV13-SC
Statistical Analysis 7: Comparison: V114-SC vs V114-IM; Injection Site Pain; Test type: Other; p = 0.333, Miettinen & Nurminen method; Difference in Percentages = 9.7, 95% CI 2-sided [-10.0 to 28.9] — Difference = % V114-SC minus % V114-IM
Statistical Analysis 8: Comparison: V114-SC vs PCV13-SC; Injection Site Pain; Test type: Other; p = 0.760, Miettinen & Nurminen method; Difference in Percentages = -3.2, 95% CI 2-sided [-23.4 to 17.2] — Difference = % V114-SC minus % PCV13-SC
Statistical Analysis 9: Comparison: V114-IM vs PCV13-SC; Injection Site Pain; Test type: Other; p = 0.205, Miettinen & Nurminen method; Difference in Percentages = -13.0, 95% CI 2-sided [-32.2 to 7.1] — Difference = % V114-IM minus % PCV13-SC
Statistical Analysis 10: Comparison: V114-SC vs V114-IM; Injection Site Swelling; Test type: Other; p = 0.128, Miettinen & Nurminen method; Difference in Percentages = 13.0, 95% CI 2-sided [-3.9 to 29.7] — Difference = % V114-SC minus % V114-IM
Statistical Analysis 11: Comparison: V114-SC vs PCV13-SC; Injection Site Swelling; Test type: Other; p = 0.779, Miettinen & Nurminen method; Difference in Percentages = -2.0, 95% CI 2-sided [-17.0 to 13.0] — Difference = % V114-SC minus % PCV13-SC
Statistical Analysis 12: Comparison: V114-IM vs PCV13-SC; Injection Site Swelling; Test type: Other; p = 0.076, Miettinen & Nurminen method; Difference in Parentages = -15.0, 95% CI 2-sided [-31.5 to 1.7] — Difference = % V114-IM minus % PCV13-SC

2. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs were decreased appetite (appetite loss), somnolence (drowsiness), irritability and urticaria (hives/welts).
Time Frame: Day 1 to Day 14 post each vaccination
Population: Analysis population consisted of all randomized participants who received at least one dose of trial vaccine.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-SC | V114-IM | PCV13-SC
Number analyzed (Participants) | 44 | 45 | 43
Percentage of Participants
  Decreased Appetite (Appetite Loss) | 25.0 | 35.6 | 34.9
  Somnolence (Drowsiness) | 70.5 | 60.0 | 74.4
  Irritability | 81.8 | 71.1 | 74.4
  Urticaria (Hives/Welts) | 9.1 | 4.4 | 7.0
Statistical Analysis 1: Comparison: V114-SC vs V114-IM; Decreased Appetite (Appetite Loss); Test type: Other; p = 0.282, Miettinen & Nurminen method; Difference in Percentages = -10.6, 95% CI 2-sided [-29.1 to 8.7] — Difference = % V114-SC minus % V114-IM
Statistical Analysis 2: Comparison: V114-SC vs PCV13-SC; Decreased Appetite (Appetite Loss); Test type: Other; p = 0.317, Miettinen & Nurminen method; Difference in Percentages = -9.9, 95% CI 2-sided [-28.7 to 9.5] — Difference= % V114-SC minus % PCV13-SC
Statistical Analysis 3: Comparison: V114-IM vs PCV13-SC; Decreased Appetite (Appetite Loss); Test type: Other; p = 0.948, Miettinen & Nurminen method; Difference in Percentages = 0.7, 95% CI 2-sided [-19.2 to 20.4] — Difference= % V114-IM minus % PCV13-SC
Statistical Analysis 4: Comparison: V114-SC vs V114-IM; Somnolence (Drowsiness); Test type: Other; p = 0.303, Miettinen & Nurminen method; Difference in Percentages = 10.5, 95% CI 2-sided [-9.4 to 29.6] — Difference = % V114-SC minus % V114-IM
Statistical Analysis 5: Comparison: V114-SC vs PCV13-SC; Somnolence (Drowsiness); Test type: Other; p = 0.681, Miettinen & Nurminen method; Difference in Percentages = -4.0, 95% CI 2-sided [-22.6 to 15.0] — Difference= % V114-SC minus % PCV13-SC
Statistical Analysis 6: Comparison: V114-IM vs PCV13-SC; Somnolence (Drowsiness); Test type: Other; p = 0.153, Miettinen & Nurminen method; Difference in Percentages = -14.4, 95% CI 2-sided [-33.2 to 5.4] — Difference= % V114-IM minus % PCV13-SC
Statistical Analysis 7: Comparison: V114-SC vs V114-IM; Irritability; Test type: Other; p = 0.237, Miettinen & Nurminen method; Difference in Percentages = 10.7, 95% CI 2-sided [-7.2 to 28.2] — Difference = % V114-SC minus % V114-IM
Statistical Analysis 8: Comparison: V114-SC vs PCV13-SC; Irritability; Test type: Other; p = 0.406, Miettinen & Nurminen method; Difference in Percentages = 7.4, 95% CI 2-sided [-10.3 to 25.0] — Difference= % V114-SC minus % PCV13-SC
Statistical Analysis 9: Comparison: V114-IM vs PCV13-SC; Irritability; Test type: Other; p = 0.729, Miettinen & Nurminen method; Difference in Percentages = -3.3, 95% CI 2-sided [-21.8 to 15.5] — Difference= % V114-IM minus % PCV13-SC
Statistical Analysis 10: Comparison: V114-SC vs V114-IM; Urticaria (Hives/Welts); Test type: Other; p = 0.385, Miettinen & Nurminen method; Difference in Percentages = 4.6, 95% CI 2-sided [-7.1 to 17.5] — Difference = % V114-SC minus % V114-IM
Statistical Analysis 11: Comparison: V114-SC vs PCV13-SC; Urticaria (Hives/Welts); Test type: Other; p = 0.719, Miettinen & Nurminen method; Difference in Percentages = 2.1, 95% CI 2-sided [-11.0 to 15.4] — Difference= % V114-SC minus % PCV13-SC
Statistical Analysis 12: Comparison: V114-IM vs PCV13-SC; Urticaria (Hives/Welts); Test type: Other; p = 0.610, Miettinen & Nurminen method; Difference in Percentages = -2.5, 95% CI 2-sided [-14.9 to 8.9] — Difference= % V114-IM minus % PCV13-SC

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event (SAE)
Description: An SAE is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine was determined by the investigator.
Time Frame: Up to 4 weeks post vaccination 4 (~14.5 months)
Population: Analysis population consisted of all randomized participants who received at least one dose of trial vaccine.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-SC | V114-IM | PCV13-SC
Number analyzed (Participants) | 44 | 45 | 43
Percentage of Participants | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants Meeting the Serotype-specific Immunoglobulin G (IgG) Threshold of ≥0.35 µg/mL
Description: Serotype-specific pneumococcal IgG antibody was measured using pneumococcal electrochemiluminescence (PnECL). The percentage of participants with serotype-specific IgG ≥0.35 µg/mL was summarized for each serotype.
Time Frame: One month post vaccination 3 (~3 months after Vaccination 1)
Population: Analysis population consisted of those participants who were not considered protocol violators.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-SC | V114-IM | PCV13-SC
Number analyzed (Participants) | 44 | 45 | 43
Percentage of Participants
  Serotype (ST) 1: number analyzed (Participants) | 44 | 45 | 42
  Serotype (ST) 1 | 100.0 | 100.0 | 100.0
  ST 3: number analyzed (Participants) | 44 | 45 | 42
  ST 3 | 100.0 | 97.8 | 100.0
  ST 4: number analyzed (Participants) | 44 | 45 | 42
  ST 4 | 100.0 | 100.0 | 100.0
  ST 5: number analyzed (Participants) | 44 | 45 | 42
  ST 5 | 100.0 | 100.0 | 100.0
  ST 6A: number analyzed (Participants) | 44 | 45 | 42
  ST 6A | 97.7 | 100.0 | 100.0
  ST 6B: number analyzed (Participants) | 44 | 45 | 42
  ST 6B | 90.9 | 93.3 | 100.0
  ST 7F: number analyzed (Participants) | 44 | 45 | 42
  ST 7F | 100.0 | 97.8 | 100.0
  ST 9V: number analyzed (Participants) | 44 | 45 | 42
  ST 9V | 100.0 | 100.0 | 100.0
  ST 14: number analyzed (Participants) | 44 | 45 | 42
  ST 14 | 97.7 | 100.0 | 100.0
  ST 18C: number analyzed (Participants) | 44 | 45 | 42
  ST 18C | 100.0 | 100.0 | 100.0
  ST 19A: number analyzed (Participants) | 44 | 45 | 42
  ST 19A | 100.0 | 100.0 | 100.0
  ST 19F: number analyzed (Participants) | 44 | 45 | 42
  ST 19F | 100.0 | 100.0 | 100.0
  ST 23F: number analyzed (Participants) | 44 | 45 | 42
  ST 23F | 97.7 | 100.0 | 97.6
  ST 22F: number analyzed (Participants) | 44 | 45 | 42
  ST 22F | 95.5 | 100.0 | 4.8
  ST 33F: number analyzed (Participants) | 44 | 45 | 42
  ST 33F | 81.8 | 88.9 | 0.0
Statistical Analysis 1: Comparison: V114-SC vs PCV13-SC; ST 1; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: V114-IM vs PCV13-SC; ST 1; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 3: Comparison: V114-SC vs V114-IM; ST 1; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 4: Comparison: V114-SC vs PCV13-SC; ST 3; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114- SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 5: Comparison: V114-IM vs PCV13-SC; ST 3; Test type: Other; Difference in Percentages = -2.2, 95% CI 2-sided [-11.7 to 6.3] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 6: Comparison: V114-SC vs V114-IM; ST 3; Test type: Other; Difference in Percentages = 2.2, 95% CI 2-sided [-6.0 to 11.6] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 7: Comparison: V114-SC vs PCV13-SC; ST 4; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference=% V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 8: Comparison: V114-IM vs PCV13-SC; ST 4; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 9: Comparison: V114-SC vs V114-IM; ST 4; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 10: Comparison: V114-SC vs PCV13-SC; ST 5; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 11: Comparison: V114-IM vs PCV13-SC; ST 5; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 12: Comparison: V114-SC vs V114-IM; ST 5; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 13: Comparison: V114-SC vs PCV13-SC; ST 6A; Test type: Other; Difference in Percentages = -2.3, 95% CI 2-sided [-11.9 to 6.3] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 14: Comparison: V114-IM vs PCV13-SC; ST 6A; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 15: Comparison: V114-SC vs V114-IM; ST 6A; Test type: Other; Difference in Percentages = -2.3, 95% CI 2-sided [-11.9 to 5.8] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 16: Comparison: V114-SC vs PCV13-SC; ST 6B; Test type: Other; Difference in Percentages = -9.1, 95% CI 2-sided [-21.2 to -0.2] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 17: Comparison: V114-IM vs PCV13-SC; ST 6B; Test type: Other; Difference in Percentages = -6.7, 95% CI 2-sided [-17.9 to 2.1] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 18: Comparison: V114-SC vs V114-IM; ST 6B; Test type: Other; Difference in Percentages = -2.4, 95% CI 2-sided [-15.6 to 10.2] — Difference=% V114 SC minus % V114 IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 19: Comparison: V114-SC vs PCV13-SC; ST 7F; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114 SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 20: Comparison: V114-IM vs PCV13-SC; ST 7F; Test type: Other; Difference in Percentages = -2.2, 95% CI 2-sided [-11.7 to 6.3] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 21: Comparison: V114-SC vs V114-IM; ST 7F; Test type: Other; Difference in Percentages = 2.2, 95% CI 2-sided [-6.0 to 11.6] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 22: Comparison: V114-SC vs PCV13-SC; ST 9V; Test type: Other; Differences in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 23: Comparison: V114-IM vs PCV13-SC; ST 9V; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 24: Comparison: V114-SC vs V114-IM; ST 9V; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 25: Comparison: V114-SC vs PCV13-SC; ST 14; Test type: Other; Difference in Percentages = -2.3, 95% CI 2-sided [-11.9 to 6.3] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 26: Comparison: V114-IM vs PCV13-SC; ST 14; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 27: Comparison: V114-SC vs V114-IM; ST 14; Test type: Other; Difference in Percentages = -2.3, 95% CI 2-sided [-11.9 to 5.8] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 28: Comparison: V114-SC vs PCV13-SC; ST 18C; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 29: Comparison: V114-IM vs PCV13-SC; ST 18C; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 30: Comparison: V114-SC vs V114-IM; ST 18C; Test type: Other; Differences in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 31: Comparison: V114-SC vs PCV13-SC; ST 19A; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference=% V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 32: Comparison: V114-IM vs PCV13-SC; ST 19A; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 33: Comparison: V114-SC vs V114-IM; ST 19A; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 34: Comparison: V114-SC vs PCV13-SC; ST 19F; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference=% V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 35: Comparison: V114-IM vs PCV13-SC; ST 19F; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 36: Comparison: V114-SC vs V114-IM; ST 19F; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 37: Comparison: V114-SC vs PCV13-SC; ST 23F; Test type: Other; Difference in Percentages = 0.1, 95% CI 2-sided [-9.8 to 10.4] — Difference=% V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 38: Comparison: V114-IM vs PCV13-SC; ST 23F; Test type: Other; Difference in Percentages = 2.4, 95% CI 2-sided [-5.7 to 12.4] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 39: Comparison: V114-SC vs V114-IM; ST 23F; Test type: Other; Difference in Percentages = -2.3, 95% CI 2-sided [-11.9 to 5.8] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 40: Comparison: V114-SC vs PCV13-SC; ST 22F; Test type: Other; Difference in Percentages = 90.7, 95% CI 2-sided [77.2 to 96.4] — Difference=% V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 41: Comparison: V114-IM vs PCV13-SC; ST 22F; Test type: Other; Difference in Percentages = 95.2, 95% CI 2-sided [84.1 to 98.7] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 42: Comparison: V114-SC vs V114-IM; ST 22F; Test type: Other; Difference in Percentages = -4.5, 95% CI 2-sided [-15.2 to 3.6] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 43: Comparison: V114-SC vs PCV13-SC; ST 33F; Test type: Other; Difference in Percentages = 81.8, 95% CI 2-sided [67.9 to 90.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 44: Comparison: V114-IM vs PCV13-SC; ST 33F; Test type: Other; Difference in Percentages = 88.9, 95% CI 2-sided [76.4 to 95.2] — Difference=% V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 45: Comparison: V114-SC vs V114-IM; ST 33F; Test type: Other; Difference in Percentages = -7.1, 95% CI 2-sided [-22.7 to 8.2] — Difference=% V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method

5. Secondary Outcome: Serotype-specific IgG Geometric Mean Concentrations (GMCs)
Description: The anti-pneumococcal polysaccharide (PnPs) serotype-specific IgG Geometric Mean Concentrations (GMCs) were determined using an electrochemiluminescence assay.
Time Frame: 1 month post vaccination 3 (~3 months after Vaccination 1)
Population: Analysis population consisted of those participants who were not considered protocol violators.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114-SC | V114-IM | PCV13-SC
Number analyzed (Participants) | 44 | 45 | 43
μg/mL
  ST 1: number analyzed (Participants) | 44 | 45 | 42
  ST 1 | 4.03 [3.33 to 4.88] | 4.55 [3.76 to 5.50] | 5.30 [4.36 to 6.45]
  ST 3: number analyzed (Participants) | 44 | 45 | 42
  ST 3 | 3.95 [3.20 to 4.89] | 4.52 [3.66 to 5.57] | 3.04 [2.44 to 3.78]
  ST 4: number analyzed (Participants) | 44 | 45 | 42
  ST 4 | 5.40 [4.63 to 6.29] | 6.02 [5.17 to 7.01] | 7.48 [6.39 to 8.75]
  ST 5: number analyzed (Participants) | 44 | 45 | 42
  ST 5 | 3.51 [2.80 to 4.40] | 3.98 [3.19 to 4.98] | 4.20 [3.33 to 5.29]
  ST 6A: number analyzed (Participants) | 44 | 45 | 42
  ST 6A | 2.09 [1.70 to 2.57] | 2.30 [1.88 to 2.82] | 3.33 [2.69 to 4.11]
  ST 6B: number analyzed (Participants) | 44 | 45 | 42
  ST 6B | 1.51 [1.14 to 1.99] | 1.72 [1.31 to 2.27] | 2.85 [2.14 to 3.78]
  ST 7F: number analyzed (Participants) | 44 | 45 | 42
  ST 7F | 2.95 [2.42 to 3.59] | 3.32 [2.73 to 4.03] | 4.85 [3.97 to 5.94]
  ST 9V: number analyzed (Participants) | 44 | 45 | 42
  ST 9V | 4.18 [3.45 to 5.06] | 4.75 [3.93 to 5.74] | 5.54 [4.55 to 6.74]
  ST 14: number analyzed (Participants) | 44 | 45 | 42
  ST 14 | 11.43 [8.99 to 14.53] | 13.79 [10.87 to 17.48] | 13.54 [10.59 to 17.31]
  ST 18C: number analyzed (Participants) | 44 | 45 | 42
  ST 18C | 3.10 [2.58 to 3.72] | 3.17 [2.64 to 3.80] | 4.48 [3.72 to 5.41]
  ST 19A: number analyzed (Participants) | 44 | 45 | 42
  ST 19A | 6.27 [5.15 to 7.63] | 5.25 [4.33 to 6.38] | 7.22 [5.90 to 8.83]
  ST 19F: number analyzed (Participants) | 44 | 45 | 42
  ST 19F | 5.42 [4.65 to 6.32] | 5.85 [5.02 to 6.80] | 7.62 [6.51 to 8.92]
  ST 23F: number analyzed (Participants) | 44 | 45 | 42
  ST 23F | 2.56 [2.04 to 3.20] | 2.57 [2.06 to 3.21] | 3.24 [2.57 to 4.07]
  ST 22F: number analyzed (Participants) | 44 | 45 | 42
  ST 22F | 6.82 [5.10 to 9.13] | 10.35 [7.76 to 13.80] | 0.05 [0.04 to 0.07]
  ST 33F: number analyzed (Participants) | 44 | 45 | 42
  ST 33F | 1.15 [0.81 to 1.62] | 1.56 [1.11 to 2.19] | 0.05 [0.03 to 0.06]
Statistical Analysis 1: Comparison: V114-SC vs PCV13-SC; ST 1; Test type: Other; Geometric Mean Concentration (GMC) Ratio = 0.76, 95% CI 2-sided [0.58 to 1.00] — GMC Ratio=GMC V114-SC/GMC PCV13-SC. Based on an analysis of variance (ANOVA) model with natural log-transformed antibody responses as response variable and vaccination group as a single factor
Statistical Analysis 2: Comparison: V114-IM vs PCV13-SC; Test type: Other; GMC Ratio = 0.86, 95% CI 2-sided [0.65 to 1.13] — GMC Ratio=GMC V114-IM/GMC PCV13-SC. Based on an ANOVA model with natural log-transformed antibody responses as response variable and vaccination group as a single factor
Statistical Analysis 3: Comparison: V114-SC vs V114-IM; Test type: Other; GMC Ratio = 0.89, 95% CI 2-sided [0.68 to 1.16] — GMC Ratio=GMC V114-SC/GMC V114-IM. Based on an ANOVA model with natural log-transformed antibody responses as response variable and vaccination group as a single factor
Statistical Analysis 4: Comparison: V114-SC vs PCV13-SC; ST 3; Test type: Other; GMC Ratio = 1.30, 95% CI 2-sided [0.96 to 1.76] — GMC Ratio=GMC V114-SC/GMC PCV13-SC. Based on an ANOVA model with natural log-transformed antibody responses as response variable and vaccination group as a single factor
Statistical Analysis 5: Comparison: V114-IM vs PCV13-SC; ST 3; Test type: Other; GMC Ratio = 1.49, 95% CI 2-sided [1.10 to 2.01] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: V114-SC vs V114-IM; ST 3; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.65 to 1.18] — GMC Ratio=GMC V114-SC/GMC V114 IM. Based on an ANOVA model with natural log-transformed antibody responses as response variable and vaccination group as a single factor
Statistical Analysis 7: Comparison: V114-SC vs PCV13-SC; ST 4; Test type: Other; GMC Ratio = 0.72, 95% CI 2-sided [0.58 to 0.90] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 8: Comparison: V114-IM vs PCV13-SC; ST 4; Test type: Other; GMC Ratio = 0.81, 95% CI 2-sided [0.65 to 1.00] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: V114-SC vs V114-IM; ST 4; Test type: Other; GMC Ratio = 0.90, 95% CI 2-sided [0.72 to 1.11] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 10: Comparison: V114-SC vs PCV13-SC; ST 5; Test type: Other; GMC Ratio = 0.84, 95% CI 2-sided [0.60 to 1.16] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 11: Comparison: V114-IM vs PCV13-SC; ST 5; Test type: Other; GMC Ratio = 0.95, 95% CI 2-sided [0.69 to 1.31] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: V114-SC vs V114-IM; ST 5; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.64 to 1.21] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 13: Comparison: V114-SC vs PCV13-SC; ST 6A; Test type: Other; GMC Ratio = 0.63, 95% CI 2-sided [0.47 to 0.84] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 14: Comparison: V114-IM vs PCV13-SC; ST 6A; Test type: Other; GMC Ratio = 0.69, 95% CI 2-sided [0.52 to 0.93] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 15: Comparison: V114-SC vs V114-IM; ST 6A; Test type: Other; GMC Ratio = 0.91, 95% CI 2-sided [0.68 to 1.21] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 16: Comparison: V114-SC vs PCV13-SC; ST 6B; Test type: Other; GMC Ratio = 0.53, 95% CI 2-sided [0.36 to 0.79] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 17: Comparison: V114-IM vs PCV13-SC; ST 6B; Test type: Other; GMC Ratio = 0.60, 95% CI 2-sided [0.41 to 0.90] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 18: Comparison: V114-SC vs V114-IM; ST 6B; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.59 to 1.30] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 19: Comparison: V114-SC vs PCV13-SC; ST 7F; Test type: Other; GMC Ratio = 0.61, 95% CI 2-sided [0.46 to 0.81] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 20: Comparison: V114-IM vs PCV13-SC; ST 7F; Test type: Other; GMC Ratio = 0.68, 95% CI 2-sided [0.52 to 0.90] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 21: Comparison: V114-SC vs V114-IM; ST 7F; Test type: Other; GMC Ratio = 0.89, 95% CI 2-sided [0.67 to 1.17] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 22: Comparison: V114-SC vs PCV13-SC; ST 9V; Test type: Other; GMC Ratio = 0.75, 95% CI 2-sided [0.57 to 0.99] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 23: Comparison: V114-IM vs PCV13-SC; ST 9V; Test type: Other; GMC Ratio = 0.86, 95% CI 2-sided [0.65 to 1.13] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 24: Comparison: V114-SC vs V114-IM; ST 9V; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.67 to 1.15] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 25: Comparison: V114-SC vs PCV13-SC; ST 14; Test type: Other; GMC Ratio = 0.84, 95% CI 2-sided [0.60 to 1.19] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 26: Comparison: V114-IM vs PCV13-SC; ST 14; Test type: Other; GMC Ratio = 1.02, 95% CI 2-sided [0.72 to 1.43] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 27: Comparison: V114-SC vs V114-IM; ST 14; Test type: Other; GMC Ratio = 0.83, 95% CI 2-sided [0.59 to 1.16] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 28: Comparison: V114-SC vs PCV13-SC; ST 18C; Test type: Other; GMC Ratio = 0.69, 95% CI 2-sided [0.53 to 0.90] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 29: Comparison: V114-IM vs PCV13-SC; ST 18C; Test type: Other; GMC Ratio = 0.71, 95% CI 2-sided [0.54 to 0.92] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 30: Comparison: V114-SC vs V114-IM; ST 18C; Test type: Other; GMC Ratio = 0.98, 95% CI 2-sided [0.76 to 1.27] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 31: Comparison: V114-SC vs PCV13-SC; ST 19A; Test type: Other; GMC Ratio = 0.87, 95% CI 2-sided [0.66 to 1.15] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 32: Comparison: V114-IM vs PCV13-SC; ST 19A; Test type: Other; GMC Ratio = 0.73, 95% CI 2-sided [0.55 to 0.96] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 33: Comparison: V114-SC vs V114-IM; ST 19A; Test type: Other; GMC Ratio = 1.19, 95% CI 2-sided [0.90 to 1.57] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 34: Comparison: V114-SC vs PCV13-SC; ST 19F; Test type: Other; GMC Ratio = 0.71, 95% CI 2-sided [0.57 to 0.89] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 35: Comparison: V114-IM vs PCV13-SC; ST 19F; Test type: Other; GMC Ratio = 0.77, 95% CI 2-sided [0.62 to 0.95] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 36: Comparison: V114-SC vs V114-IM; ST 19F; Test type: Other; GMC Ratio = 0.93, 95% CI 2-sided [0.75 to 1.15] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 37: Comparison: V114-SC vs PCV13-SC; ST 23F; Test type: Other; GMC Ratio = 0.79, 95% CI 2-sided [0.57 to 1.09] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 38: Comparison: V114-IM vs PCV13-SC; ST 23F; Test type: Other; GMC Ratio = 0.80, 95% CI 2-sided [0.58 to 1.09] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 39: Comparison: V114-SC vs V114-IM; ST 23F; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.73 to 1.36] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 40: Comparison: V114-SC vs PCV13-SC; ST 22F; Test type: Other; GMC Ratio = 134.88, 95% CI 2-sided [88.91 to 204.62] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 41: Comparison: V114-IM vs PCV13-SC; ST 22F; Test type: Other; GMC Ratio = 204.60, 95% CI 2-sided [135.18 to 309.69] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 42: Comparison: V114-SC vs V114-IM; ST 22F; Test type: Other; GMC Ratio = 0.66, 95% CI 2-sided [0.44 to 0.99] — [estimate comment as in outcome 5, analysis 6]
Statistical Analysis 43: Comparison: V114-SC vs PCV13-SC; ST 33F; Test type: Other; GMC Ratio = 25.11, 95% CI 2-sided [15.34 to 41.13] — [estimate comment as in outcome 5, analysis 4]
Statistical Analysis 44: Comparison: V114-IM vs PCV13-SC; ST 33F; Test type: Other; GMC Ratio = 34.18, 95% CI 2-sided [20.93 to 55.83] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 45: Comparison: V114-SC vs V114-IM; ST 33F; Test type: Other; GMC Ratio = 0.73, 95% CI 2-sided [0.45 to 1.19] — [estimate comment as in outcome 5, analysis 6]

6. Secondary Outcome: Percentage of Participants Meeting Threshold Values for Protective Responses to DTaP-IPV (Diphtheria Toxin, Tetanus Toxin, Pertussis Toxin, Pertussis Filamentous Hemagglutinin (FHA) and Polio Virus Type 1/2/3)
Description: DTaP-IPV antibody titers were measured by neutralization assay (diphtheria toxin and poliovirus 1/2/3), particle agglutination assay (tetanus toxin) and enzyme-linked immunosorbent assay (ELISA) methodology (pertussis PT and pertussis FHA) 1 month post vaccination 3. Threshold values were: Diphtheria toxin level ≥0.1 IU/mL, Pertussis PT level ≥10 EU/mL, Pertussis FHA level ≥10 EU/mL, Tetanus toxin level ≥0.01 IU/mL, Neutralizing antibody (NA) titers of Polio virus types 1/2/3 ≥1:8.
Time Frame: 1 month post vaccination 3 (~3 months after Vaccination 1)
Population: Analysis population consisted of those participants who were not considered protocol violators.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-SC | V114-IM | PCV13-SC
Number analyzed (Participants) | 44 | 45 | 43
Percentage of Participants
  Diphtheria toxin | 97.7 | 95.6 | 95.2
  Tetanus toxin | 100.0 | 100.0 | 97.6
  Pertussis toxin | 100.0 | 100.0 | 100.0
  Pertussis FHA | 100.0 | 100.0 | 100.0
  Poliovirus Type 1 | 100.0 | 100.0 | 100.0
  Poliovirus Type 2 | 100.0 | 100.0 | 100.0
  Poliovirus Type 3 | 100.0 | 100.0 | 100.0
Statistical Analysis 1: Comparison: V114-SC vs PCV13-SC; Diphtheria Toxin; Test type: Other; Difference in Percentages = 2.5, 95% CI 2-sided [-7.7 to 13.9] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: V114-IM vs PCV13-SC; Diphtheria Toxin; Test type: Other; Difference in Percentages = 0.3, 95% CI 2-sided [-10.8 to 12.0] — Difference = % V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 3: Comparison: V114-SC vs V114-IM; Diphtheria Toxin; Test type: Other; Difference in Percentages = 2.2, 95% CI 2-sided [-8.0 to 13.0] — Difference = % V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 4: Comparison: V114-SC vs PCV13-SC; Tetanus Toxin; Test type: Other; Difference in Percentages = 2.4, 95% CI 2-sided [-5.8 to 12.4] — Difference = % V114 SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 5: Comparison: V114-IM vs PCV13-SC; Tetanus Toxin; Test type: Other; Difference in Percentages = 2.4, 95% CI 2-sided [-5.7 to 12.4] — Difference = % V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 6: Comparison: V114-SC vs V114-IM; Tetanus Toxin; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference = % V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 7: Comparison: V114-SC vs PCV13-SC; Pertussis Toxin; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 8: Comparison: V114-IM vs PCV13-SC; Pertussis Toxin; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference = % V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 9: Comparison: V114-SC vs V114-IM; Pertussis Toxin; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference = % V114 SC minus % V114 IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 10: Comparison: V114-SC vs PCV13-SC; Pertussis FHA; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 11: Comparison: V114-IM vs PCV13-SC; Pertussis FHA; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference = % V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 12: Comparison: V114-SC vs V114-IM; Pertussis FHA; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference = % V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 13: Comparison: V114-SC vs PCV13-SC; Poliovirus Type 1; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 14: Comparison: V114-IM vs PCV13-SC; Poliovirus Type 1; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference = % V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 15: Comparison: V114-SC vs V114-IM; Poliovirus Type 1; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference = % V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 16: Comparison: V114-SC vs PCV13-SC; Poliovirus Type 2; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 17: Comparison: V114-IM vs PCV13-SC; Poliovirus Type 2; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference = % V114-IM minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 18: Comparison: V114-SC vs V114-IM; Poliovirus Type 2; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference = % V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 19: Comparison: V114-SC vs PCV13-SC; Poliovirus Type 3; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 8.5] — Difference = % V114-SC minus % PCV13-SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 20: Comparison: V114-IM vs PCV13-SC; Poliovirus Type 3; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-7.9 to 8.5] — Difference = % V114-IM minus % PCV13 -SC. The 95% CI is based on the Miettinen and Nurminen method
Statistical Analysis 21: Comparison: V114-SC vs V114-IM; Poliovirus Type 3; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-8.1 to 7.9] — Difference = % V114-SC minus % V114-IM. The 95% CI is based on the Miettinen and Nurminen method

ADVERSE EVENTS:
Time Frame: Non-serious AEs: up to 14 days post each vaccination SAEs and All-cause Mortality: up to 4 weeks post vaccination 4 (~14.5 months)
Arm/Group | V114-SC | V114-IM | PCV13-SC
All-Cause Mortality (participants affected / at risk) | 0/44 | 1/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/44 | 3/45 | 2/43
Other Adverse Events (participants affected / at risk) | 44/44 | 44/45 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114-SC (N=44) | V114-IM (N=45) | PCV13-SC (N=43)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114-SC (N=44) | V114-IM (N=45) | PCV13-SC (N=43)
Constipation (Gastrointestinal disorders) | 1 (6) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (8) | 6 (6)
Injection site erythema (General disorders) | 44 (236) | 37 (145) | 41 (217)
Injection site induration (General disorders) | 40 (215) | 35 (144) | 43 (229)
Injection site pain (General disorders) | 17 (43) | 13 (30) | 18 (49)
Injection site swelling (General disorders) | 38 (174) | 33 (87) | 38 (163)
Injection site warmth (General disorders) | 3 (10) | 2 (4) | 6 (10)
Pyrexia (General disorders) | 27 (63) | 25 (50) | 27 (53)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 11 (19) | 16 (30) | 15 (32)
Somnolence (Nervous system disorders) | 31 (64) | 27 (75) | 32 (81)
Irritability (Psychiatric disorders) | 36 (90) | 32 (87) | 32 (102)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 8 (8) | 9 (11)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1) | 1 (1)
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (3) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03848065/Prot_SAP_000.pdf